CLINICAL TRIAL: NCT07357766
Title: A Placebo-controlled Comparability Study to Compare Two Presentations of CagriSema in Participants With Overweight or Obesity
Brief Title: A Research Study to Compare Different Versions of Injectable CagriSema and Placebo in People With Excess Body Weight
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-8166; U1111-1317-0133 (Other: World Health Organization); 2024-520448-41 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2026-01-21; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CagriSema B in device 2 + Placebo in device 1 (Experimental): Participants will receive CagriSema B in device 2 followed by placebo matched to CagriSema in device 1 subcutaneously once weekly in a dose escalation manner for 16 weeks until the target maintenance dose and further continue to receive the same dose for up to 44 weeks.
  Interventions: Drug: Cagrisema
- CagriSema in device 1 + Placebo in device 2 (Experimental): Participants will receive CagriSema in device 1 followed by placebo matched to CagriSema B in device 2 subcutaneously once weekly in a dose escalation manner for 16 weeks until the target maintenance dose and further continue to receive the same dose for up to 44 weeks.
  Interventions: Drug: Cagrisema
- Placebo in device 1 + Placebo in device 2 (Placebo Comparator): Participants will receive placebo matched to Cagrisema in device 1 followed by placebo matched to CagriSema B in device 2 subcutaneously once weekly for up to 44 weeks.
  Interventions: Drug: Placebo CagriSema

INTERVENTIONS:
Drug: Cagrisema — Cagrisema (Cagrilintide and Semaglutide) will be administered subcutaneously using device 1 or device 2.
  Arms: CagriSema B in device 2 + Placebo in device 1; CagriSema in device 1 + Placebo in device 2
Drug: Placebo CagriSema — Placebo matched to Cagrilintide and Placebo matched to Semaglutide will be administered subcutaneously using device 1 or device 2.
  Arms: Placebo in device 1 + Placebo in device 2

SUMMARY:
This study is being done to find out how well a medicine called CagriSema helps people with overweight or obesity lose weight. CagriSema is still being tested in studies and is not yet available for doctors to prescribe. In this study the sponsor will compare two version of CagriSema injected by two different types of injection devices. Which treatment participants get is decided by chance using a computer program, so neither participants nor study staff will know which treatment is given. The study will last for about one year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (sex at birth)
* Age 18 years or above at the time of signing the informing consent.
* Body Mass Index (BMI) is greater than or equal to (>= ) 30.0 kilograms per square metre (kg/m^2) or BMI >= 27.0 kg/m^2 with the presence of at least one obesity-related complication including, but not limited to, hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease.

Exclusion Criteria:

* Glycosylated haemoglobin (HbA1c) >= 6.5 % (48 millimoles per mole [mmol/mol]) as measured by the central laboratory at screening.
* History of type 1 or type 2 diabetes.
* Previous exposure to CagriSema in a clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2026-06-09 (Estimated); Primary Completion 2027-11-16 (Estimated); Study Completion 2028-01-04 (Estimated)

PRIMARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to end of treatment (week 44)
  Measured in percentage (%).

SECONDARY OUTCOMES:
Number of TEAEs (treatment emergent adverse events) | From baseline (week 0) to end of study (week 51)
  Measured in count of events.
Number of TESAEs (Treatment emergent serious adverse events) | From baseline (week 0) to end of study (week 51)
  Measured in count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (96):
- United States (7):
  - Cahaba Research, Pelham, Alabama
  - ForCare Clinical Research, Tampa, Florida
  - Arcturus HC PLC Troy Med Res, Troy, Michigan
  - Palm Research Center Inc., Las Vegas, Nevada
  - Alliance for Multispecialty Research, Norman, Oklahoma
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Capital Clin Res Ctr,LLC, Olympia, Washington
- Bulgaria (13):
  - IPSMC - Dr. Nikolay Kostadinov EOOD, Burgas
  - Medical Center Viva Feniks OOD, Dobrich
  - IPSOMC Dr. Miglena Rizova Ltd., Kyustendil
  - UMHAT Pulmed, Endocrinology and Metabolic Diseases, Plovdiv
  - UMHAT Sveti Georgi EAD, Plovdiv, Clinic of Endocrinology, Plovdiv
  - MHAT Sveta Karidad EAD, Plovdiv
  - DCC Iztok EOOD, Plovdiv
  - Medical Centre Razgrad OOD, Razgrad
  - DCC VII - Sofia EOOD, Endocrinology, Sofia
  - Diagnostic-Consultative Anti-Aging and Rejuvenation Center Hill Clinic EAD, Sofia
  - Medical Center Medical Plus EOOD, Varna
  - DCC Mladost - M Varna OOD, Varna
  - AIPSMC Dr. Artin Magardichyan EOOD, Varna
- Denmark (3):
  - Sanos Clinic - Gandrup, Gandrup
  - Sanos Clinic - Vejle, Vejle
  - Regionshospitalet Viborg - Karkirurgisk Afsnit, Viborg
- Greece (7):
  - 251 Air Force General Hospital - Department of Endocrinology & Diabetes, Athens
  - General Hospital Of Athens G Gennimatas - Department of Endocrinology, Athens
  - Laiko General Hospital Of Athens - A' Propaedeutic Clinic of Internal Medicine-Diabetes Centre, Athens
  - Athens Medical Center S.A. (Iatriko Athinon) - Diabetes and Obesity Unit, Marousi
  - Athens Medical Center S.A. (Iatriko P. Falirou) - Diabetes and Clinical Research Center, Palaió Fáliro
  - General Hospital Of Thessaloniki G Gennimatas - Internal Medicine Clinic, Thessaloniki
  - Thermi Clinic S.A. - Diabetes and Internal Medicine Department, Thessaloniki
- Hungary (6):
  - Arina Trial Research Kft., Orosháza, Bekes County
  - Belinus Bt., Debrecen, Hajdú-Bihar
  - Debreceni Egyetem, Debrecen, Hajdú-Bihar
  - Borbánya Praxis E.Ü. Kft., Nyíregyháza, Szabolcs-Szatmar Varmegye
  - ClinDiab Egészségügyi Szolgáltató és Kereskedelmi Kft., Budapest
  - Szegedi Tudományegyetem, Szeged
- Malaysia (11):
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Seri Manjung, Seri Manjung, Perak
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Miri, Miri, Sarawak
  - Klinik Kesihatan Kuang, Rawang, Selangor
  - University Technology MARA (UiTM) - Sg Buloh, Sungai Buloh, Selangor
  - Klinik Kesihatan Kuala Kedah, Kuala Kedah
  - Hospital Melaka, Malacca
  - Hospital Queen Elizabeth II, Sabak Bernam
- Poland (11):
  - Gabinet Leczenia Otylosci i Chorob Dietozaleznych, Bialystok
  - Centrum Medyczne Kermed Renata Bijata-Bronisz I Ewa Kowalinska Sp. j., Bydgoszcz
  - Niepubliczny Zakład Opieki Zdrowotnej BIF-MED S.C. Arkadiusz Wawiernia, Mariola Roykiewicz, Rafał Roykiewicz, Bytom
  - NZOZ Mediart Centrum Zdrowia Matarnia, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - ID Clinic Arkadiusz Pisula, Mysłowice
  - Clinical Best Solutions Sp. z o.o., Sp. k, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Kardio Life - Tomasz Borkowski, Włocławek
  - Velocity Nova Sp. z o.o., Zamość
  - Prywatna Praktyka Lekarska Anna Chudoba, Żyrardów
- Portugal (6):
  - ULS De Braga, E.P.E. - Hospital de Braga, Braga
  - ULS Do Alto Ave, E.P.E. - Hospital Senhora da Oliveira - Guimarães, Guimarães
  - Hospital S. Francisco, S.A, Leiria
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - Affidea Montijo - UCardio, Montijo
  - Cardiolima Centro Diagnostico Cardio-Pulmonar De Ponte De Lima Lda, Ponte de Lima
- Romania (7):
  - Thera Card S.R.L, Brasov
  - Kilostop Junior SRL, Bucharest
  - SC Diamed Obesity SRL, Galati
  - Arcadia Policlinic SRL, Iași
  - Spital Judetean De Urgenta Satu Mare, Satu Mare
  - SC Gensan SRL, Policlinica ASTRA, Sibiu
  - Spitalul Clinic Judetean De Urgenta Targu Mures, Târgu Mureş
- Slovakia (5):
  - MED-CENTRUM, s.r.o., Martin
  - KARDIOMED NZ, s.r.o., Nové Zámky
  - SVAJDLEROVA, s.r.o., Prešov
  - ENRIN, s.r.o., Rimavská Sobota
  - DIAB s.r.o., Rožňava
- South Africa (6):
  - Soweto Clinical Trial Centre, Johannesburg, Gauteng
  - Ezintsha Research Centre, Johannesburg, Gauteng
  - Shop#1 Health Emporium, Midrand, Gauteng
  - Dr Vawda's site, Durban, KwaZulu-Natal
  - Dr T Padayachee, Durban, KwaZulu-Natal
  - Dr Moosa's Rooms, Gauteng, Lenasia
- Switzerland (4):
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital Olten, Olten
  - Stoffwechselzentrum St. Gallen, Sankt Gallen
  - Diabetes Adipositas Zentrum Zürich, Zollikerberg
- Taiwan (4):
  - Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City
  - Kuang Tien General Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - Taipei Municipal Wan Fang Hospital_Division of Endocrinology & Metabolism, Taipei
- Thailand (6):
  - Hat Yai hospital, Hat Yai, Changwat Songkhla
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai, Chiang Mai
  - RIHES-CMU_Research Institute for Health Sciences, Chiang Mai
  - Thammasat Hospital_CRC, Pathum Thani

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisktrials.com
URL: https://novonordisk-trials.com